CLINICAL TRIAL: NCT06684015
Title: The Effect of Intrathecal Morphine and Erector Spina Plan Block on Serum Cytokine Levels and Chronic Pain in Caesarean Section Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Fatih Kurt, Research Assistant, Ankara University
Other Study IDs: İ02-121-24
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Cesarean Delivery; Postoperative Pain; Cytokine Levels; Chronic Pain, Postoperative
Keywords: intrathecal morphine; cesarean delivery; acute postoperative pain; spinal anesthesia; tumor necrosis factor alpha; interleukin 6; interleukin 10; Chronic pain, postoperative; erector spinae plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples With DNA — In order to evaluate the basal serum cytokine levels from each patient, 5 milliliters (ml) of venous blood will be taken before the operation (after monitoring-before spinal anesthesia). In order to evaluate the changes in serum cytokine levels after the operation, the moment when the first blood sample is taken will be considered as the beginning; 5 ml venous blood samples will be taken at the 6th and 24th hours. The collected venous blood samples will be transferred in a biochemistry tube containing separator gel in accordance with the blood product transfer protocol, and the serum samples obtained will be stored at -80 degrees after being centrifuged for 10 minutes at 3000G in the biochemistry laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intratechal morphine: Addition of intrathecal morphine as an adjuvant to local anesthesia in routine spinal anesthesia application and multimodal analgesia applications
  Interventions: Drug: İNTRATECHAL MORPHİNE GROUP
- Erector spinae plane block: Application of erector spinae plane block and multimodal analgesia applications at the end of the operation after routine spinal anesthesia application
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Drug: İNTRATECHAL MORPHİNE GROUP — Addition of intrathecal morphine as an adjuvant to local anesthesia in routine spinal anesthesia application and multimodal analgesia applications
  Groups: Intratechal morphine
Procedure: Erector Spinae Plane Block — Application of erector spinae plane block and multimodal analgesia applications at the end of the operation after routine spinal anesthesia application
  Groups: Erector spinae plane block

SUMMARY:
Working Title The Effect of Intrathecal Morphine and Erector Spina Plan Block on Serum Cytokine Levels and Chronic Pain in Caesarean Section Surgery

Study Description This study aims to evaluate the effects of intrathecal morphine added as an adjuvant to local anesthesia during spinal anesthesia and the erector spinae plane block applied at the end of cesarean surgery on postoperative serum cytokine levels, pain intensity, need for rescue analgesia, hospital anxiety and depression levels, quality of obstetric recovery, and the development of chronic postoperative pain.

Study Type Study Design: Observational Model: Two parallel groups Time Perspective: Prospective

Interventions Intervention Type: Drug and Block Procedure Details: In patients included in the study, intrathecal morphine is administered as an adjuvant to local anesthesia during spinal anesthesia first group. At the end of surgery, an erector spinae plane block is performed other group.

Primary Outcome Measures Serum Cytokine Levels Time Frame: 0., 6. and 24. Hours Assessment Method: Serum biochemical analyses

Pain Intensity and Need for Rescue Analgesia Time Frame: 2., 4., 6., 12. and 24. hours, assessed using the Numeric Rating Scale(NRS)

Hospital Anxiety and Depression Levels Time Frame: Preoperative and at 24 hours postoperatively Assessment Method: Hospital Anxiety and Depression Scale (HADS)

Quality of Obstetric Recovery Score Time Frame: At 24 hours postoperatively

Chronic Postoperative Pain Development Time Frame: Evaluated at 4 months postoperatively Assessment Method: Short Form McGill Pain Questionnaire-2

DETAILED DESCRIPTION:
-Design of the Study The study was designed as observational, prospective, two parallel groups and single-blind. The study planned to investigate the effects of intrathecal morphine and erector spinae plane block application on serum cytokine levels and chronic pain in cesarean surgery. In order to evaluate the inflammatory response caused by surgical stress at the cytokine level and to investigate the effects of this response on acute postoperative and chronic pain, patient demographic information, medical data, biological material to be collected and volunteer surveys will be analyzed and evaluated.

Both methods to be applied are routinely used methods in cesarean surgery anesthesia applications as part of the multimodal analgesia method.

In our study, where the volunteer population of pregnant patients planned to undergo elective cesarean surgery was formed at the Gynecology and Obstetrics Clinic of Ankara University Faculty of Medicine, it is thought that the number of volunteers meeting the inclusion criteria will be reached in approximately 4 months with the evaluation of the retrospective patient population. The follow-up period of the patients included in the study was 3 months, and the total period for the study was planned as 7 months if the targeted number of patients could be reached.

Volunteers may exercise their right to withdraw from the study at any stage of the study without giving any reason. Volunteers included in the study but in cases of unsuccessful spinal anesthesia application, need for repeat spinal anesthesia application, removal of early intraoperative spinal block, application of sedation, conversion to general anesthesia, development of surgical complications (bleeding, atony, etc.), hemodynamic instability, development of need for blood product transfusion, etc. will be excluded from the study and their routine perioperative care will continue.

-Study groups Morphine group: Addition of intrathecal morphine as an adjuvant to local anesthesia in routine spinal anesthesia application and multimodal analgesia applications Erector spinae plane block group: Application of erector spinae plane block and multimodal analgesia applications at the end of the operation after routine spinal anesthesia application

Hyperbaric bupivacaine calculated at an appropriate dose of 0.5% concentration will be applied to the patients in spinal anesthesia application. The maximum dose of intrathecal hyperbaric bupivacaine has been stated as 18 milligrams (mg) (21).

The methods routinely applied to each patient for multimodal analgesia; 1 g paracetamol (max 4 g/day), 50 mg dexketoprofen (max 150 mg/day) and 8 mg dexamethasone (max 16 mg/kg) will be applied to all patients intravenously (IV) following umbilical cord clamping. Paracetamol will continue to be administered as 1 gram every 8 hours in the postoperative period. The doses to be applied are within the safe range for each drug.

During our clinical practice, 50-100 micrograms (mcg) of morphine can be added as an adjuvant agent when spinal anesthesia is routinely applied. In this study, patients who were administered 50 mcg of morphine intrathecally will be included in the study as it is less associated with side effects such as postoperative nausea, vomiting, urinary retention, etc. (21). Erector spinae plane block is applied to patients who have undergone spinal anesthesia, in addition, at the end of the operation, at the level of the 9th thoracic vertebra, under ultrasound guidance, bilaterally, with a volume of 20 milliliters (ml) of 0.25% bupivacaine solution for each side, with a total bupivacaine dose of 100 mg. In this study, observational data on these patients will be collected. The complication rate associated with erector spinae plane block can be seen as low as 2 cases in 10,000 patients (22).

- Taking and preserving blood samples and studying cytokine (Interleukin-6, Tumor Necrosis Factor-alpha, Interleukin-10) levels A 5-milliliter (ml) venous blood sample will be taken from each patient before the operation (after monitoring-before spinal anesthesia) in order to evaluate the basal serum cytokine levels. In order to evaluate the changes in serum cytokine levels after the operation, the moment the first blood sample is taken is considered as the beginning; 5 ml venous blood samples will be taken at 6 and 24 hours. The half-life of Interleukin-6 is known to be <1 hour (23), the half-life of TNF-alpha is 6 minutes (24), and the half-life of Interleukin-10 is approximately 1 hour (25). Although many time periods are stated in the literature for the purpose of controlling cytokine levels (6, 11, 12), the hours planned for taking control blood samples were determined as 6 and 24 hours, considering the onset and end times of the effects of the methods used in the study arms.

The venous blood samples taken will be transferred in a biochemistry tube containing separator gel in accordance with the blood product transfer protocol and centrifuged for 10 minutes at 3000G in the biochemistry laboratory, and the serum samples obtained will be stored at -80 degrees. When the targeted number of patients is reached, serum cytokine levels will be studied with ELISA (Enzyme-Linked ImmunoSorbent Assay) kits and the results will be recorded. After all the samples are collected, the serums will be studied collectively by Assoc. Prof. Dr. Özlem Doğan in the Cebeci Central Biochemistry Laboratory of Ankara University Faculty of Medicine.

- Anesthesia applications Patients will be evaluated by the anesthesiologist for routine preoperative examination, information and obtaining their consent before the operation. The consents of patients who accept regional anesthesia/analgesia applications and volunteering in the study will be obtained by answering all their questions and providing detailed information. Each patient taken to the operation room; Standard monitoring with electrocardiography (ECG), non-invasive blood pressure (NIBP) and pulse oximetry (SpO2) will be applied. Intravenous (IV) access will be provided with an 18 gauge (G) intracatheter.

All patients included in the study will receive spinal anesthesia for anesthesia.

Following the blood collection procedure, patients will be positioned for spinal anesthesia and hydration will be initiated with isolene-S with a target volume of 15 ml/kg. After aseptic conditions are provided in the sitting position, the intervals of the lumbar 4th and 5th vertebrae (L4-L5) spinous processes will be palpated and a 26G Quincke-type spinal needle will be inserted from the midline and the appropriate dose of medication will be administered after the cerebrospinal fluid (CSF) flow is observed. In spinal anesthesia application to patients in the morphine arm, 50 mcg morphine (Double dilution method (26); 10 milligram (mg) / ml morphine ampoule is diluted with 9 ml of 0.9% NaCl. 9 ml of the resulting 1 mg/ml mixture is discarded and the remaining 1 ml is diluted with 9 ml of 0.9% NaCl. 0.5 ml of the resulting morphine/isotonic mixture with a concentration of 100 mcg/ml is drawn into the calculated bupivacaine syringe) will be added as an adjuvant to local anesthesia. After the procedure, patients will be placed in a supine position on their left side at 15 degrees, and oxygenation will be provided with a mask if necessary. Sensory block will be checked with pinprick test and cold-hot discrimination. The operation will be started after the targeted block level is achieved at the 4th-6th thoracic dermatome (T4-T6) level. The block level will be checked every 15 minutes (min) during the operation. In case of unsuccessful spinal anesthesia, repetition of spinal anesthesia, or conversion of anesthesia to general anesthesia due to intraoperative spinal anesthesia insufficiency, patients will be excluded from the study and their routine follow-up and care will continue. Vital signs of the patients will be monitored during the operation. A decrease in mean blood pressure (MBP) to more than 20% of the baseline value or systolic blood pressure (SBP) to below 90 mmHg will be considered hypotension and 100 mcg ephedrine will be administered IV. A decrease in heart rate below 50 beats/min will be considered bradycardia and 0.5 mg atropine will be administered IV.

If there are no contraindications, all patients will be administered 1 gram (gr)cefazolin, 8 mg ondansetron, 40 mg pantoprazole and 10 IU oxytocin as a slow infusion IV following umbilical cord clamping, and 0.2 mg methylergonovine will be administered intramuscularly (IM).

In all patients included in the study, if there is no contraindication for multimodal analgesia, IV 1 gr paracetamol, 50 mg dexketoprofen and 8 mg dexamethasone will be routinely administered following umbilical cord clamping.

Only local anesthetic drugs are administered to patients in the erector spinae plane block arm during spinal anesthesia. Patients in this arm will be placed in the lateral decubitus position with the assistance of 2 assistants at the end of the operation, and the transverse process of the T12 vertebra and the 12th rib will be imaged with ultrasound (USG) and the transverse process of the T9 vertebra will be determined by counting in the cranial direction. Under aseptic conditions, the block needle (21G, 100 mm) will be advanced under the erector spinae muscle and 2-3 ml of 0.9% physiological serum and 20 ml of 0.25% bupivacaine will be administered after hydrodissection and interfascial drug spread will be observed. The procedure will be repeated for the other side.

At the end of the operation, all patients included in the study will be transferred to the postoperative recovery unit (PODU). Patients without additional problems will be transferred from the PODU to their rooms and their postoperative follow-up will be performed.

1 g of paracetamol will be administered to the patients IV once every 8 hours for postoperative analgesia. Patients with a numerical ratio scale-11 (NRS-11) value of 4 and above will be administered 75 mg diclofenac (maximum dose 150 mg/day) IM as rescue analgesia.

-Data to be recorded perioperatively The time the patients arrive at the table for the operation, the time the spinal anesthesia is applied, the number of spinal anesthesia attempts, the time the sensory block reaches the T4 level, the operation start time, the baby's exit time, the operation end time and the patient's exit time after the operation, the amount of medication used for spinal anesthesia, the Bromage score when the block reaches the T4 dermatome, the amount of fluid given to the patient intraoperatively and the amount of urine the patient produces and the baby's 1st and 5th minute APGAR values will be recorded.

The severity of the patients' surgically developed pain at rest/motion and with coughing, the presence and severity of back and headache, the severity of nausea and vomiting, their satisfaction levels, their breastfeeding status, their vital values and whether they need additional analgesics and if so, the time and amount will be recorded.

Following the first blood sample, control blood samples will be taken at the 6th and 24th hours.

Hospital Anxiety and Depression Scale Before the operation and 24 hours after the operation; in order to evaluate hospital anxiety and depression levels and to compare the effects of the applied methods on these data, the "Hospital Anxiety and Depression Scale" questionnaire will be applied to the volunteers included in the study a total of 2 times.

Obstetric Recovery Quality Score (ObsQoR-11) At 24 hours after the operation; in order to evaluate the effect of the applied methods on the quality of recovery after surgery, the "Obstetric Recovery Quality Score (ObsQoR-11)" questionnaire will be applied to the volunteers included in the study a total of 1 time.

Short Form McGill Pain Questionnaire-2 In order to evaluate the effects of the applied methods on the development of chronic pain after surgery in the 4th month after the operation, the "Short Form McGill Pain Questionnaire-2" questionnaire will be applied to the volunteers included in the study a total of 1 time via telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* ASA II
* Elective surgery
* Spinal anesthesia
* To accept participation in the study and regional anesthesia applications

Exclusion Criteria:

* Under 18 years old
* BMI (body mass index) >35 kilograms/meter2 (kg/m2)
* ASA III and above
* Multiple pregnancy
* Previous abdominal surgery
* History of malignancy
* Contraindication for regional anesthesia
* Known history of allergy to the drugs to be used
* Presence of chronic pain (migraine, fibromyalgia, etc.)
* History of substance abuse
* Regular use of painkillers (simple analgesics, gabapentinoids, opioids)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In our study, healthy pregnant patients who were planned to undergo elective cesarean section in Ankara University Faculty of Medicine, Department of Obstetrics and Gynecology constituted the volunteer population.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
postoperative serum cytokine | 24 hours
  We aimed to investigate the effects of intrathecal morphine administered as adjuvant in spiral anesthesia and erector spina plan block performed at the end of the operation on postoperative serum cytokine (Interleukin-6, Tumor Necrosis Factor-alpha, Interleukin-10) levels.
  In order to evaluate the basal serum cytokine levels from each patient, 5 milliliters (ml) of venous blood will be taken before the operation (after monitoring-before spinal anesthesia). In order to evaluate the changes in serum cytokine levels after the operation, the moment when the first blood sample is taken will be considered as the beginning; 5 ml of venous blood will be taken at the 6th and 24th hours. Although many time periods are stated in the literature for the control of cytokine levels (6, 11, 12), the hours planned for the control blood samples were determined as the 6th and 24th hours, considering the start and end times of the effects of the methods used in the study arms.
Chronic pain | 4 months
  We aimed to investigate the effects of intrathecal morphine administered as adjuvant in spiral anesthesia and erector spina plan block performed at the end of the operation on chronic pain in patients undergoing cesarean section surgery.
  The assessment will be made with the McGill Short Form Pain Questionnaire-2. The questionnaire consists of 22 items. Each question is evaluated with a Numeric Rating Scale. A low score is associated with less pain, while a high score is associated with more pain.

SECONDARY OUTCOMES:
postoperative acute pain | 24 hours
  To investigate the effects of intrathecal morphine administered as adjuvant in spinal anesthesia and erector spina plan block performed at the end of the operation on postoperative acute pain in patients undergoing cesarean section surgery.
  Acute pain will be assessed postoperatively with a Numeric rating scale at 2, 4, 6, 12 and 24 hours.
  A low score is associated with less pain and a high score is associated with more pain.
amount of additional analgesic rescue | 24 hours
  To investigate the effects of intrathecal morphine administered as adjuvant in spinal anesthesia and erector spina plan block performed at the end of the operation on amount of additional analgesic rescue in patients undergoing cesarean section surgery.
  During the postoperative follow-up, if the pain status of the patients is NRS>4, IM NSAII will be applied as an additional analgesic. It will be evaluated whether there is a difference between the groups in terms of rescue analgesics.
Hospital anxiety and depression | 24 hours
  To investigate the effects of intrathecal morphine administered as adjuvant in spinal anesthesia and erector spina plan block performed at the end of the operation on patient anxiety in patients undergoing cesarean section surgery.
  The preoperative and postoperative conditions of the patients will be evaluated with the Hospital Anxiety and Depression Scale applied in the preoperative period and at the 24th hour postoperatively.
  Lower scores in the scale assessment are associated with lower anxiety and depression.
Obstetric Quality of Recovery | 24 hours
  To investigate the effects of intrathecal morphine administered as adjuvant in spinal anesthesia and erector spina plan block performed at the end of the operation on quality of recovery in patients undergoing cesarean section surgery.
  Patients will be assessed at 24 hours with the Obstetric Recovery Quality score. A higher score is associated with increased recovery quality.

CONTACTS AND LOCATIONS:
Overall Officials: Suheyla Karadag Erkoc, Associate Professor, Principal Investigator — Ankara University Faculty of Medicine
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I haven't decided yet.